CLINICAL TRIAL: NCT00555113
Title: Evolution of Visual Impairment During Pseudoxanthoma Elasticum
Status: Completed | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Other Study IDs: 2
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-11

CONDITIONS: Pseudoxanthoma Elasticum
Keywords: pseudoxanthoma elasticum; Visual acuity; Choroidal neovascularization; angioid streaks
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Choroidal Neovascularization; Angioid Streaks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: pseudoxanthoma elasticum

SUMMARY:
Pseudoxanthoma elasticum is a disease whom frequency is estimated about 1/50000 to 1/100 000. There is a female preponderance with a sex-ratio of 2:1. PXE is transmitted according either to an autosomal dominant mode or to an autosomal recessive one. Mutations in the ABCC6 gene on chromosome 16p13.1 have recently been identified causing PXE. The elastic fibers slowly become mineralized mainly in the skin, the eyes, and the cardiovascular system. PXE is a multisystem disease that includes a spectrum of clinical manifestations affecting the skin, the eye or the cardiovascular system as well as other tissues. It can be responsible for severe and life threatening complications. Skin changes are usually the first manifestations and begin in early childhood. The vital prognosis of PXE depends on the severity of the cardiovascular lesions that could be responsible for sudden death in children and young adults.

Ocular manifestations are quite constant and include chorioretinal scarring, pigmentary changes or angioid streaks. The natural evolution of the angioid streaks leads to their enlargement or to the occurrence of subfoveal choroidal neovascularizations and hemorrhages leaving macular scares. A self-monitoring is recommended since early treatment of subfoveal CNV is the only way to minimize their pejorative consequences. The gold standard treatment of the CNV consists in the photocoagulation. New therapeutics has been developed including photodynamic therapy or intravitreal injection of anti-angiogenic agents and they seems to be effective to reduce the immediate complications of a limited CNV. This evolution explains that 50 to 70 % of the patients have a poor vision or legal blindness of one or both eyes. However, little is known about the age of occurrence of visual impairment in PXE patients. That is the reason why we decided to review the ophthalmologic status and visual history of our population of PXE patients according to their age.

DETAILED DESCRIPTION:
A retrospective review of all cases of PXE patients referred by the Department of Genetics should be performed. This ophthalmologic examination has been conducted as part of the usual follow up for such PXE patients or for the needs of a treatment of complications of angioid streaks such as CNV complications.

As we studied the age of poor vision occurrence, we propose to take in account the first examination when a best-corrected visual acuity (BCVA) under 20/50 was observed. All past medical events obtains from the data of the patients will be recorded, especially ophthalmologic ones.

ELIGIBILITY:
Inclusion Criteria:

* pseudoxanthoma elasticum confirmed by the Department of Genetics according to the usual clinical, histological or genetic criterion.

Exclusion Criteria:

* No pseudoxanthoma elasticum

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with pseudoxanthoma elasticum confirmed by the Department of Genetics according to the usual clinical, histological or genetic criterion.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2000-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Visual acuity according to age | 7 years

SECONDARY OUTCOMES:
Macular aspect and outcoming of choroidal neovascularization | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Christophe ORSSAUD, MD, Principal Investigator — department of ophthalmology, HEGP, AP - HP, France
Locations (1):
- Department of ophthalmology, HEGP, Paris, Paris, France

REFERENCES:
- [Background] Pakalnis L, Makoroto J. Reproduction and the test tube baby. Can Nurse. 1977 Feb;73(2):34-8. PMID 264800